CLINICAL TRIAL: NCT05407688
Title: Compatibility of Participation Levels of Adolescents With Attention Deficit and Hyperactivity Disorder in Terms of Adolescent and Parent Perspectives
Brief Title: Compatibility of Participation Levels of Adolescents With Attention Deficit and Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof., Akdeniz University
Other Study IDs: 2021/339
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: attention deficit hyperactivity disorder; adolescent; participation; PEM-CY
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD group: Adolescents with ADHD
- Health group: Adolescents without ADHD

SUMMARY:
The goal of this study is to assess the agreement between the outcomes of adolescents with attention deficit hyperactivity disorder (ADHD) who participated in Participation and Environment Measurement Child & Youth (PEM-CY) by the adolescent and primary caregiver. There are a few studies in the literature that look at the participation of teenagers with ADHD, but none that look at the participation of adolescents with ADHD from both the perspective of the adolescents and the primary caregivers. The primary caregiver's measurement results and the adolescents' measurements do not concur, according to this study's hypothesis.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is one of the most common neurodevelopmental disorders in childhood. In addition to fundamental symptoms like inattention and hyperactivity/impulsivity, ADHD can be accompanied by a variety of diseases. Adolescents with ADHD are less likely to participate in activities at home, school, or in the community as a result of this. In comparison to children without ADHD, Shimoni et al. found that children with ADHD participate less frequently in most leisure activities, like formal leisure activities less, and have a lower desire for participation in specific leisure activities, such as physical and social leisure activities.

Adolescents and their primary caregivers have disagreements on a variety of topics. This disagreement is also likely to arise when it comes to choose who will participate. Furthermore, while measuring the level of engagement, the need of gathering information from various sources is clear. The Participation and Environment Measurement-Children and Youth (PEM-CY) is a scale that evaluates parents' or caregivers' involvement with children and young people in the home, school, and community. Adolescents with ADHD had lower levels of participation in the home, school, and community than control groups, according to research. However, no study analyzing this level of bidirectional participation could be found in the existing literature (adolescent-primary caregivers).

As a result, the primary goal of this study is to examine the participation of adolescents with ADHD from the perspectives of adolescents and primary caregivers using The Participation and Environment Measure for Children and Youth (PEM-CY), as well as to demonstrate the agreement between these two evaluations. Furthermore, it will be compared to healthy controls in terms of participation and agreement rates.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 years and 12 years;
* Diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) by a child and adolescent health psychiatrist, regardless of subtype, according to DSM-V criteria
* Have cognitive ability to follow instructions for assessment measures

Exclusion Criteria:

* Children have any other psychiatric diagnosis like autism spectrum disorder, psychotic symptoms, depression, etc.
* Children have any neurological or orthopedic disorders like head injury, cerebral palsy, epileptic seizure, visual and speech disorder.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents with ADHD at 12-17 years old and their parents. Healthy adolescents at aged 7-12 years old and their parents.
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of participation | baseline
  Participation and Environment Measurement Child & Youth (PEM-CY) is a parent-report questionnaire to assess participation and environment factors in the home, at school, and within community settings. The participation sections included 10 activities in the home setting, five activities in the school setting and 10 in the community setting. For each activity, parents are asked to determine the participation frequency (how frequently has the child participates with eight options: daily to never), participation involvement (how involved the child is while participating in the activity rated on a five-point scale: very involved to minimally involved) and whether change is desired (do the parents want to see change in the child's participation in this type of activity: no or yes, with five different types of change).

SECONDARY OUTCOMES:
Evaluation of ADHD symptoms | Baseline
  The Conners' Ratin Scale - Revised (CRS-R) was designed to address the need for a multimodal assessment of children and adolescents' behavioral difficulties and contains a parent form, a teacher form, and an adolescent self report form. The parent form, the CPRS-R, is appropriate for use with parents of children and adolescents ages 3 through 17. The Long Form contains 80 items and can be completed by most parents/guardians in approximately 20 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klassen AF, Miller A, Fine S. Agreement between parent and child report of quality of life in children with attention-deficit/hyperactivity disorder. Child Care Health Dev. 2006 Jul;32(4):397-406. doi: 10.1111/j.1365-2214.2006.00609.x. PMID 16784495
- [Result] Dada S, Andersson AK, May A, Andersson EE, Granlund M, Huus K. Agreement between participation ratings of children with intellectual disabilities and their primary caregivers. Res Dev Disabil. 2020 Sep;104:103715. doi: 10.1016/j.ridd.2020.103715. Epub 2020 Jun 20. PMID 32574934
- [Result] Kaya Kara O, Turker D, Kara K, Yardimci-Lokmanoglu BN. Psychometric properties of the Turkish version of Participation and Environment Measure for Children and Youth. Child Care Health Dev. 2020 Nov;46(6):711-722. doi: 10.1111/cch.12801. Epub 2020 Aug 19. PMID 32776565
- [Result] Shimoni M, Engel-Yeger B, Tirosh E. Participation in leisure activities among boys with attention deficit hyperactivity disorder. Res Dev Disabil. 2010 Nov-Dec;31(6):1234-9. doi: 10.1016/j.ridd.2010.07.022. Epub 2010 Aug 12. PMID 20705424
- See also: Diagnostic and statistical manual of mental disorders (DSM-5®) — http://psychiatry.org/psychiatrists/practice/dsm